CLINICAL TRIAL: NCT06794827
Title: Evaluating Clinical Practice of Early Access Avacopan Treatment for ANCA-associated Vasculitis in European Countries
Brief Title: Early-access Avacopan in Real-world ANCA-associated Vasculitis
Acronym: AVAC-EUR
Status: Recruiting | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Collaborators: University of Udine (Other); University of Modena and Reggio Emilia (Other); Hospital Universitari de Bellvitge (Other); ZOL Hospital Genk Belgium (Unknown)
Responsible Party: Principal Investigator, Y.K.Onno Teng, Clinical Professor, Leiden University Medical Center
Other Study IDs: IIS-AVA-2023-0005
Record Dates: First submitted 2024-03-01; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: ANCA Associated Vasculitis
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The current study proposal aims to investigate the clinical practice variation of the initial use of avacopan for AAV patients in Europe. The study will describe patient characteristics and organ-specific clinical benefit of avacopan treatment in a unique, first-experience cohort of AAV patients. By studying the clinical practice variation of first-experience avacopan treatment, this study will be uniquely positioned to identify pivotal issues on the real-life implementation of avacopan treatment. These observational data can ultimately serve to address current knowledge gaps on avacopan treatment in AAV patients, improve the care and drug-access for AAV patients with avacopan treatment and generate new areas of research.

DETAILED DESCRIPTION:
Objective: Analyse the clinical practice variation of the early access use of avacopan in real-world treated patients with ANCA-associated vasculitis.

Study design: Observational cohort study Study population: AAV patients treated with avacopan.

Main study parameters/endpoints:

* Describe physician's treatment indications for starting avacopan
* Describe AAV patients clinical characteristics
* Describe the concomitant treatment strategies employed with avacopan
* Describe clinical outcomes of avacopan treatment
* Investigate determinants of clinical benefit as well as non-response and/or relapse within the study cohort

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of GPA or MPA
* Treatment (initiation) with avacopan
* Informed consent for use of medical data

Exclusion Criteria:

* If there is no AAV disease activity present that can be supported by an objectifiable clinical measure or assessment
* If a subject is below 16 years old

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A multicenter, non-interventional, longitudinal cohort study which will collect incident as well as prevalent AAV patients treated with an avacopan-based regimen. The cohort will include retrospective and prospective data capture on real-life management and outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Assess physician's treatment indications for starting avacopan as reported in the database questionnaire | 1 year
  Assess physician's treatment indications for starting avacopan as reported in the database questionnaire.
  Options to choose are: Refractory disease, Relapsing disease, Steroid dependent, Steroid toxicity or Other
Assess AAV patients' clinical characteristics at baseline as reported in the database questionnaire | 1 year
  Assess AAV patients' clinical characteristics at baseline as reported in the database questionnaire including:
  Gender (Male/Female) Age Date of AAV diagnosis Type AAV (GPA or MPA) Autoantibodies (PR3 or MPO) Organs affected
Assess concomitant immunosuppressive treatment strategies employed with avacopan as registered in the database questionnaire | 1 year
  Assess concomitant treatment strategies employed with avacopan at baseline, 1 month, 3 months, 6 months, 9 months, 12 months, 18 months and 24 monhts.
  Possible options include steroids, cyclophosphamide, rituximab, azathioprine or other
Assess the relevant clinical benefit of avacopan treatment at the individual patient level based on the BVAS score [0-63] | 2 years
  Assess the relevant clinical benefit of avacopan treatment at the individual patient level based on the BVAS score [0-63] as reported at baseline, 1 month, 3 months, 6 months, 9 months, 12 months, 18 months and 24 monhts.

SECONDARY OUTCOMES:
Investigate determinants of non-response and/or relapse upon avacopan treatment based on baseline characteristics registered in the database questionnaire | 2 years
  Investigate determinants of non-response and/or relapse upon avacopan treatment based on baseline characteristics registered in the database questionnaire including:
  Gender (Male/Female) Age Date of AAV diagnosis Type AAV (GPA or MPA) Autoantibodies (PR3 or MPO) Organs affected

CONTACTS AND LOCATIONS:
Overall Officials: Y.K. Onno Teng, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided